CLINICAL TRIAL: NCT01113814
Title: Performance of Acoustic Radiation Force Impulse-Imaging in Comparison to Transient Elastography for the Non-invasive Staging of Liver Fibrosis in Patients With Chronic Hepatitis C
Brief Title: Acoustic Radiation Force Impulse-Imaging in Comparison to Transient Elastography for Liver Fibrosis Staging in HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Vermehren, MD, Johann Wolfgang Goethe University Hospital
Purpose: Diagnostic
Other Study IDs: JWGUHMED1-003
Record Dates: First submitted 2010-04-27; First posted 2010-04-30 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FibroScan
Device: Acoustic Radiation Force Impulse (ARFI)- Imaging

SUMMARY:
This study will evaluate the effectiveness of Acoustic Radiation Force Impulse (ARFI)- Imaging compared to Transient Elastography (FibroScan) in differentiating liver fibrosis in patients with chronic hepatitis C. Patients who are scheduled to have a liver biopsy will also undergo ARFI and FibroScan testing. The liver biopsy will be used as the reference method. The target sample size is 433.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-79 years old
* Written consent
* Chronic Hepatitis C infection
* Liver biopsy planned or performed within the last six months
* In addition, 10 patients/center with proven liver cirrhosis without present liver biopsy can be included

Exclusion Criteria:

* Consuming illness (HIV infection, malignoma)
* Comorbidities associated to HCV (HBV, NASH, hemochromatosis, primary sclerosing cholangitis, primary biliary cirrhosis
* Antiviral therapy between liver biopsy and study inclusion
* Pacemaker or heart defibrillator
* Pregnancy or lactation
* Liver transplantation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Non-inferiority of AUROCs of Acoustic Radiation Force Impulse (ARFI)- Imaging to Transient Elastography (Fibroscan) for assessment of liver fibrosis in patients with chronic hepatitis C using liver biopsy as the reference standard.
  The diagnostic accuracy measured with the Area under the ROC curve (AUROC) is calculated for Acoustic Radiation Force Impulse (ARFI)- Imaging and Transient Elastography (Fibroscan) using histology obtained by liver biopsy as reference method in patients infected with chronic hepatitis C. The ROC curve represents sensitivity versus 1-specificity for all possible cut-off values for prediction of the different fibrosis stages, respectively. The areas under the curves (AUROC) as well as 95 % CI of AUROC are calculated.

SECONDARY OUTCOMES:
Comparison of AUROC of ARFI-Imaging and Transient Elastography with FibroMax (liver fibrosis marker)
Comparison of AUROC of ARFI and Transient Elastography with the European Liver Fibrosis-Group Marker (ELF)
Evaluation of a combination of non-invasive methods for optimising AUROC for the assessment of liver fibrosis
Evaluation of factors associated with measurement failure of ARFI-Imaging and Transient Elastography
Assessment of center variability of results

CONTACTS AND LOCATIONS:
Locations (9):
- Bordeaux University Hospital, Bordeaux, France
- Germany (7):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum der J.W. Goethe-Universität, Frankfurt am Main
  - Institut für Interdisziplinäre Medizin, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Ludwig-Maximilians-Universität-Campus Großhadern, München
- Erasmus Medical Center, Rotterdam, Netherlands